CLINICAL TRIAL: NCT07377773
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of QLS12010 Capsules in Adult Participants With Moderate-to-Severe Rheumatoid Arthritis
Brief Title: QLS12010 in Participants With Moderate-to-severe Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS12010-203
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLS12010 Capsule Dose 1 Group (Experimental)
  Interventions: Drug: QLS12010
- QLS12010 Capsule Dose 2 Group (Experimental)
  Interventions: Drug: QLS12010
- QLS12010 Capsule Dose 3 Group (Experimental)
  Interventions: Drug: QLS12010
- Placebo Group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: QLS12010 — QLS12010 oral capsule
  Arms: QLS12010 Capsule Dose 1 Group; QLS12010 Capsule Dose 2 Group; QLS12010 Capsule Dose 3 Group
Drug: placebo — Matching placebo oral capsule
  Arms: Placebo Group

SUMMARY:
The objective of this randomized, double-blind, placebo-controlled phase II clinical trial is to investigate the safety and efficacy of QLS12010 in subjects with moderate-to-severe rheumatoid arthritis.The main questions it aims to answer are:

• Efficacy and safety of QLS12010 in participants with rheumatoid arthritis.

Participants will be randomly allocated to four treatment groups at a 1:1:1:1 ratio to compare the efficacy and safety of different dosages of QLS12010 Capsules against the placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old (inclusive).
* Diagnosed with rheumatoid arthritis as defined by the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for at least 12 weeks prior to screening; ACR functional class I-III.
* Tender joint count (TJC) ≥ 4/68 and swollen joint count (SJC) ≥ 4/66.
* High Sensitivity C-Reactive Protein (hsCRP) > Upper Limit of Normal (ULN) or erythrocyte sedimentation rate (ESR) ≥ 28 mm/h at screening.
* Inadequate response to at least one conventional synthetic disease-modifying antirheumatic drug (csDMARD) and one biologic disease-modifying antirheumatic drug (bDMARD)/ targeted synthetic disease-modifying antirheumatic drug (tsDMARD).
* Glucocorticoid dose ≤ 10 mg/day prednisone-equivalent, stable for ≥ 2 weeks pre-screening and ≥ 4 weeks pre-baseline.
* Nonsteroidal Antiinflammatory Drugs (NSAIDs) or acetaminophen, stable for ≥ 1 week pre-screening and ≥ 2 weeks pre-baseline.

Exclusion Criteria:

* Participants with other inflammatory arthritis, systemic inflammatory diseases, or Felty syndrome.
* Participants with a history of malignancy within 5 years prior to screening.
* Concurrent conditions predisposing to QT interval prolongation; QTc interval (Fridericia-corrected) > 450 ms; or thyroid-stimulating hormone (TSH) > 5 mIU/L.
* Participants with untreated recurrent migraine.
* Participants with a history of opportunistic infection within 6 months prior to ICF signing; any infection requiring hospitalization or IV anti-infective therapy within 3 months; or any acute systemic infection within 2 weeks prior to baseline.
* Participants with HIV, HBV, HCV, Treponema pallidum, or active tuberculosis (TB).
* Participants with a history of major surgery performed within 2 months prior to baseline.
* Participants with a history of severe allergic reactions or known allergy to any component of the study drug.
* Prior receipt of cell therapy (e.g., CAR-T) or T-cell engager therapy.
* Participants with a history of strong CYP3A4 inhibitors/inducers, narrow therapeutic index CYP3A substrates, strong P-gp/BCRP inhibitors, P-gp/BCRP substrates, or any QT-prolonging drugs within 4 weeks or 5 half-lives prior to baseline.
* Participants with a history of addictive drug abuse within 1 year prior to ICF signing; or alcohol abuse within 6 months prior to ICF signing.
* Participants with blood pressure > 160/100 mmHg at baseline.
* Pregnant or lactating women.
* Participants with blood donation or total blood loss ≥ 400 mL within 3 months prior to ICF signing.
* Vaccination with or exposure to live/attenuated live vaccines within 4 weeks prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2028-03-05 (Estimated); Study Completion 2028-06-05 (Estimated)

PRIMARY OUTCOMES:
Change in Disease Activity Score-C-Reactive Protein (DAS28-CRP) from Baseline at Week 12. | 12 weeks
  The DAS28-CRP score measures how active rheumatoid arthritis is. A score of 2.6 or lower indicates disease remission, while a greater score indicates more severe disease.

IPD SHARING:
Plan to Share IPD: No